CLINICAL TRIAL: NCT01193673
Title: Discovering the Gene(s) Causing Developmental Dysplasia of the Hip
Brief Title: Discovering the Gene(s) Causing Developmental Dysplasia of the Hip (DDH)
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Peters, M.D., University of Utah
Other Study IDs: 35439
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA samples are kept
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the study is to find the gene(s) responsible for causing DDH. The secondary objective of the study is to determine the mode of genetic transmission of DDH.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH), formerly known as Congenital Dislocation of the Hip (CDH) is a relatively common disorder that can lead to early onset arthritis of the hip. It is believed that DDH is the major cause of arthritis of the hip in young patients. The majority of patients with DDH are unaware of their condition. Only a very small number of these patients with the extremely severe form of the disease (dislocated hip) are identified at birth. The remaining patients usually seek help when severe arthritis is present and joint preservation treatment is not possible. The exact etiology of this condition remains elusive. Based on reports in the literature, DDH is believed to have a genetic basis.

Dr. Javad Parvizi at Rothman Institute (RT) in Philadelphia has extensive experience with this condition because their center provides joint preservation procedures such as pelvic and femoral osteotomy. They also have extensive experience with hip replacement in these patients. They are aware of some families with many affected individuals. Close history taking and examination of these patients has suggested that there may indeed be a genetic basis for DDH. Based on our findings so far, we believe that a dominant pattern of inheritance may exist, implying that this disorder may be inherited in a Mendelian manner (Single gene disorder).

Furthermore, Dr. Parvizi's group have documented a peculiar pattern of dominant inheritance in which all affected males give rise to only affected female children, suggesting that the disorder may be inherited as an X-linked dominant trait. X-linked dominant is the mode of inheritance in which a gene on the X chromosome is dominant. The X-linked dominant inheritance may in part account for the large number of females affected with the trait. Understanding the inheritance mechanism of this disease will allow better genetic counseling and monitoring of affected individuals and their families.

The reason behind this study is to investigate the possible genetic inheritance of the disease. Knowing this information will allow us to test patients for the disease early and before arthritis develops. In addition it is possible that better treatments may be designed based on this knowledge.

DDH is a relatively common condition. Although the most severe form of DDH is usually diagnosed during birth (dislocated hip), the majority (>80%) of patients with this condition do not even know that they suffer from this disease and usually discover their condition when disabling arthritis of the hip develops in early adulthood.

ELIGIBILITY:
Inclusion Criteria:

* All patients with radiographic and clinical diagnosis of DDH will be included.

Exclusion Criteria:

* Other forms of arthritis:
* osteoarthritis
* inflammatory arthropathies
* vascular necrosis

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with hip dysplasia and their family members.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-01; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Analyze whole exome sequencing for causative mutation(s) in Fibrodysplasia Ossificans Progressiva (FOP) and other genetic variations. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Peters, MD, Principal Investigator — University of Utah Orthopaedic Center
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States